CLINICAL TRIAL: NCT07126600
Title: A Data Collection Study for Echocardiography-Based Software Assessment
Brief Title: Data Collection for Echocardiography-Based Software Assessment
Status: Completed | Type: Observational
Sponsor: Anumana, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DOC-2499
Record Dates: First submitted 2025-07-28; First posted 2025-08-17 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation; Left Atrial Appendage Closure; Cardiovascular Diseases
MeSH Terms: conditions — Atrial Fibrillation; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- LAAC Patient Cohort: Participants undergoing standard-of-care imaging as part of a left atrial appendage closure (LAAC) procedure. Data will be collected prospectively for software validation purposes.
  Interventions: Other: No investigational intervention administered

INTERVENTIONS:
Other: No investigational intervention administered — No investigational intervention administered

SUMMARY:
This is a prospective, observational study collecting data from routine clinical care. The information gathered will be used to support the evaluation of a software-based tool. No investigational procedures or treatments are introduced, and all data are obtained as part of standard-of-care activities.

DETAILED DESCRIPTION:
This is a prospective, observational study designed to collect data from routine clinical procedures related to a specific cardiac intervention. Data will be collected from multiple sites and compiled into a centralized dataset. The dataset will be used to support the evaluation of software-based tools intended to assist in clinical decision-making.

No investigational interventions are introduced as part of the study, and all activities align with standard-of-care practices at participating institutions. The study may also support future analyses related to the performance and usability of the software.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing a standard left atrial appendage closure procedure with associated imaging.

Exclusion Criteria:

* Did not provide authorization to use data for research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing a standard cardiac procedure as part of routine clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-07-11 (Actual); Primary Completion 2025-11-19 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
Comparison of Imaging-Derived Measurements | At the time of imaging assessment (single study visit)
  Comparison of left atrial appendage measurements (millimeters) from two imaging modalities against a CT-based reference standard.

CONTACTS AND LOCATIONS:
Overall Officials: Leon Ptaszek, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (6):
- United States (6):
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Southcoast Hospital, New Bedford, Massachusetts
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - University of Buffalo, Amherst, New York
  - Montefiore Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No